CLINICAL TRIAL: NCT00327405
Title: A Retrospective Study of Surgical Outcomes.
Brief Title: Results of Ocular Compression and Suture Release in Trabeculectomy and Combined Surgery
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Other Study IDs: UCJSC001
Record Dates: First submitted 2006-05-17; First posted 2006-05-18 (Estimated); Last update posted 2006-05-18 (Estimated); Status verified 2006-01

CONDITIONS: Primary Open Angle Glaucoma
Keywords: POAG; Primary Open Angle Glaucoma; Trabeculectomy; Combined Phacotrabeculectomy; Combined Glaucoma Cataract Surgery; Releasable Suture; Ocular Compresssion
MeSH Terms: conditions — Glaucoma, Open-Angle

SUMMARY:
The use of ocular compression and suture release have helped to improve the safety and decrease the risks of glaucoma filtering surgery. This study looks at the decrease in intraocular pressure and glaucoma medications required following glaucoma filtering surgery.

DETAILED DESCRIPTION:
A retrospective review of surgical results in eyes with at least six months followup was performed for trabeculectomy and combined phacoemulsification-trabeculectomy surgery. A total of 141 eyes were studied.

ELIGIBILITY:
Inclusion Criteria:

* Primary Open Angle Glaucoma
* Six Months Followup
* No previous surgery

Exclusion Criteria:

* Less Than Six Months Followup
* Previous glaucoma surgery

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: John S Cohen, MD, Principal Investigator — University of Cincinnati Department of Ophthalmology
Locations (1):
- Cincinnati Eye Institute, Cincinnati, Ohio, United States